CLINICAL TRIAL: NCT00784927
Title: A Phase 2 Study of Lenalidomide, Rituximab, Cyclophosphamide and Dexamethasone (LR-CD) for Untreated Low Grade Non-Hodgkin Lymphoma Requiring Therapy
Brief Title: Lenalidomide, Rituximab, Cyclophosphamide, and Dexamethasone in Treating Patients With Previously Untreated Low-Grade Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0882; P30CA015083 (NIH); MC0882 (Other: Mayo Clinic Cancer Center); RV-NHL-PI-0336 (Other: Celgene Protocol); 08-001485 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-11-01; First posted 2008-11-04 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma
Keywords: stage I grade 1 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage I small lymphocytic lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage I marginal zone lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Cyclophosphamide; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Participants with symptomatic untreated low grade NHL will be treated according to a 28 day schedule for up to a maximum of 12 consecutive cycles:
  375 mg/m^2 Rituximab IV on day 1. 20 mg Lenalidomide taken orally on days 1-21. 250 mg/m^2 Cyclophosphamide orally on days 1, 8, 15. 40 mg Dexamethasone orally on days 1, 8, 15, 22.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: dexamethasone; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: dexamethasone
Drug: lenalidomide

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with rituximab, cyclophosphamide, and dexamethasone may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving lenalidomide together with rituximab, cyclophosphamide, and dexamethasone works in treating patients with previously untreated low-grade non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess tumor response to lenalidomide, rituximab, cyclophosphamide, and dexamethasone in patients with symptomatic previously untreated low-grade non-Hodgkin lymphoma.

Secondary

* To describe the adverse event profile of this regimen.
* To evaluate overall survival, progression-free survival, duration of response, and time to treatment failure associated with this regimen.
* To estimate tumor response to lenalidomide, rituximab, cyclophosphamide and dexamethasone in the subgroup of patients with lymphoplasmacytic lymphoma (Waldenstrom's macroglobulinemia).

OUTLINE: This is a multicenter study.

Patients receive oral lenalidomide once daily on days 1-21, rituximab IV on day 1, oral cyclophosphamide once daily on days 1, 8, and 15, and oral dexamethasone once daily on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed symptomatic non-Hodgkin lymphoma by biopsy within the past 6 months

  * Any of the following subtypes allowed:

    * Grade 1 or 2 lymphoma
    * Small lymphocytic lymphoma
    * Marginal zone lymphoma
    * Lymphoplasmacytic lymphoma (Waldenstrom macroglobulinemia [WM])
* Previously untreated disease that, in the investigator's opinion, requires treatment
* Measurable disease by CT or MRI scans with lymph nodes ≥ 2.0 cm in ≥ 1 dimension

  * WM patients without lymphadenopathy must meet the following criteria:

    * More than 10% lymphocytes, lymphoplasmacytic cells, or plasma cells on a bone marrow aspirate/biopsy
    * Quantitative Immunoglobulin M ≥ 400 mg/dL NOTE: A new classification scheme for adult non-Hodgkin lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,400/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2.0 mg/dL
* Total or direct bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2 times upper limit of normal (ULN) (5 times ULN if hepatic metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception at least 28 days prior to, during, and for 28 days after completion of study therapy
* Able to take acetylsalicylic acid (ASA) 325 mg/day as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin)
* No known hypersensitivity to thalidomide
* No development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No myocardial infarction within the past 6 months
* No other active malignancy requiring treatment, except for localized nonmelanomatous skin cancer or any cancer that, in the judgement of the investigator, has been treated with curative intent and will not interfere with the study treatment plan and response assessment
* No co-morbid systemic illnesses or other severe concurrent disease which, in the judgement of the investigator, would make the patient inappropriate for entry into the study or would interfere significantly with the proper assessment of safety and toxicity of study treatment
* No known positivity for HIV or infectious hepatitis A, B, or C
* No serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent
* Willing to return to Mayo Clinic enrolling institution for follow up
* Registered into the RevAssist® program and willing and able to comply with the requirements of RevAssist®

PRIOR CONCURRENT THERAPY:

* No prior lenalidomide
* No prior irradiation to ≥ 25% of the bone marrow
* More than 28 days since prior experimental drug or therapy
* No concurrent radiotherapy, chemotherapy, or immunotherapy
* No other concurrent anticancer agents or treatments, including thalidomide or investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-11; Primary Completion 2013-10 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig B Reeder, MD, Study Chair — Mayo Clinic; Thomas E. Witzig, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 36
Completed | 33
Not Completed | 3
Not completed — Cancel Prior to Initiating Treatment | 1
Not completed — Protocol Violation | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 68 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Tumor Response
Description: The proportion of responses was determined by counting the number of complete responses and partial responses and dividing by the number of evaluable patients.
  Complete Response (CR): Disappearance of all evidence of disease and disease-related symptoms. The spleen and/or liver, if considered enlarged before therapy on the basis of a physical examination or CT scan, should not be palpable on physical examination and should be considered normal size by imaging studies, and nodules related to lymphoma should disappear. If the bone marrow was involved by lymphoma before treatment, the infiltrate must have cleared on repeat bone marrow biopsy.
  Partial Response (PR): At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. No increase should be observed in the size of other nodes, liver, or spleen. No new sites of disease should be observed.
Time Frame: Up to 1 year from registration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 33
percentage of participants
  Complete Response (CR) | 30.3 [15.6 to 48.7]
  Partial Response (PR) | 54.5 [36.4 to 71.9]

2. Secondary Outcome: Tumor Response to Lenalidomide, Rituximab, Cyclophosphamide and Dexamethasone in the Subgroup of Patients With Lymphoplasmacytic Lymphoma (Waldenstrom's Macroglobulinemia).
Description: The proportion of responses in Waldenstrom's macroglobulinemia was determined by counting the number of complete responses and partial responses and dividing by the number of evaluable patients.
  Complete Response (CR): Disappearance of all evidence of disease and disease-related symptoms. The spleen and/or liver, if considered enlarged before therapy on the basis of a physical examination or CT scan, should not be palpable on physical examination and should be considered normal size by imaging studies, and nodules related to lymphoma should disappear. If the bone marrow was involved by lymphoma before treatment, the infiltrate must have cleared on repeat bone marrow biopsy.
  Partial Response (PR): At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. No increase should be observed in the size of other nodes, liver, or spleen. No new sites of disease should be observed.
Time Frame: Up to 1 year from registration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment: Participants with lymphoplasmacytic lymphoma (Waldenstrom's macroglobulinemia) will be treated according to a 28 day schedule for up to a maximum of 12 consecutive cycles and analyzed as a separate cohort:
  375 mg/m^2 Rituximab IV on day 1. 20 mg Lenalidomide taken orally on days 1-21. 250 mg/m^2 Cyclophosphamide orally on days 1, 8, 15. 40 mg Dexamethasone orally on days 1, 8, 15, 22.
  rituximab
  cyclophosphamide
  dexamethasone
  lenalidomide
Arm/Group | Treatment
Number analyzed (Participants) | 15
percentage of participants
  Complete Response (CR) | 6.7 [0.2 to 32]
  Partial Response (PR) | 66.7 [38.4 to 88.2]

3. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 1 year from registration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 33
months | NA [NA to NA] — The median overall survival time and the upper and lower confidence limits were not reached.

4. Secondary Outcome: Progression-free Survival Time
Description: Progression-free survival time is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had disease progression at the time of their death.
  Progressive disease is defined as having one of the following:
  * The appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size.
  * At least a 50% increase from nadir in the sum of the product of the dimension (SPD) of any previously involved nodes.
  * At least a 50% increase in the longest diameter of any single previously identified node more than 1 cm in its short axis.
Time Frame: Up to 1 year from registration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 33
months | 38.3 [25.2 to NA] — The 95% upper confidence limit was not reached.

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal. The distribution of time to treatment failure will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 1 year from registration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 33
months | NA [NA to NA] — The median time to treatment failure and the upper and lower confidence limits were not reached.

ADVERSE EVENTS:
Groups:
- Treatment: 40 mg Dexamethasone orally on days 1, 8, 15, 22.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 15/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=33)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3)
Vascular disorder (Vascular disorders) | 1 (1)
Sudden Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=33)
Hemoglobin decreased (Blood and lymphatic system disorders) | 28 (174)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (22)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (31)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 15 (59)
Fatigue (General disorders) | 33 (217)
Fever (General disorders) | 1 (2)
Cytokine release syndrome (Immune system disorders) | 4 (5)
Hypersensitivity (Immune system disorders) | 2 (2)
Immune system disorder (Immune system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (6)
Tooth infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 2 (3)
Leukocyte count decreased (Investigations) | 26 (109)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 28 (121)
Platelet count decreased (Investigations) | 22 (134)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 14 (36)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (52)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (3)
Cystitis (Renal and urinary disorders) | 4 (9)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 14 (34)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes